CLINICAL TRIAL: NCT01722500
Title: International Study of Childhood Obesity, Lifestyle and the Environment (ISCOLE)
Brief Title: International Study of Childhood Obesity, Lifestyle and the Environment
Acronym: ISCOLE
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: The Coca-Cola Company (Industry)
Responsible Party: Principal Investigator, Peter T. Katzmarzyk, Associate Executive Director of Population Science, Pennington Biomedical Research Center
Other Study IDs: PBRC 10042CC
Record Dates: First submitted 2012-10-29; First posted 2012-11-07 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Childhood Obesity
Keywords: International; Childhood; Obesity; ISCOLE; Pennington Biomedical Research Center; PBRC; longitudinal; multinational
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 10 year old children: 500 children with mean age 10.5 years from each of 12 countries

SUMMARY:
The primary aim of the International Study of Childhood Obesity, Lifestyle and the Environment (ISCOLE) is to determine the relationship between lifestyle characteristics and obesity in a large multi-national study of 10 year-old children, and to investigate the influence of behavioral settings and physical, social and policy environments on the observed relationships within each country.

DETAILED DESCRIPTION:
Data will be collected in 12 countries (500 children per site) from five major regions of the world (Eurasia & Africa, Europe, Latin America, North America, and the Pacific). Cross-sectional evaluations will be undertaken in each country. The physical characteristics of the children will be directly measured in order to classify their body weight and adiposity status, and physical activity and dietary patterns will be measured with the most objective techniques currently available. A concise set of environmental measures that are feasible, valid and meaningful across the international settings included in this research will also be employed. The results of this study will provide a robust examination of the correlates of obesity and weight gain in children, focusing on both sides of the energy balance equation. The results will also provide important new information that will inform the development of lifestyle interventions to address childhood obesity that can be culturally adapted for implementation around the world.

ELIGIBILITY:
Inclusion Criteria:

* students 10 years of age

Exclusion Criteria:

* has pacemaker or other internal medical devices

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: boys and girls who are approximately 10 years
Sampling Method: Non-Probability Sample
Enrollment: 7806 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Testing of Children | Baseline
  BMI (kg/m2)
Testing of Children | Baseline
  Waist Circumference (cm)
Testing of Children | Baseline
  Percent Body Fat (%)

SECONDARY OUTCOMES:
Testing of Children | Baseline
  Physical activity (minutes/day)
Testing of Children | Baseline
  Dietary intake (principal components analysis score)

CONTACTS AND LOCATIONS:
Overall Officials: Peter T. Katzmarzyk, PhD, FACSM, Principal Investigator — Pennington Biomedical Research Center; Timothy S. Church, MD, MPH, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (12):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States
- School of Health Sciences at University of South Australia, Adelaide, Australia
- Centro de Estudos do Laboratório de Aptidão Física de São Caetano do Sul (CELAFISCS), São Paulo, Brazil
- Department of Pediatrics, University of Ottawa, Ottawa, Ontario, Canada
- Tianjin Women's & Children's Health Center, Tianjin, China
- Department of Public Health School of Medicine at Universidad de los Andes, Carrera, Bogata, Colombia
- Department of Food & Environmental Sciences, University of Helsinki, Helsinki, Finland
- St John's National Academy of Health Sciences, Bangalore, Karnataka, India
- Department of Exercise, Recreation and Sports Science at Kenyatta University, Nairobi, Kenya
- Faculty of Sport Sciences and Physical Education - University of Porto, Porto, Portugal
- University of Cape Town, Rondebosch, Cape Town, South Africa
- Department of Health at University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Katzmarzyk PT, Barreira TV, Broyles ST, Champagne CM, Chaput JP, Fogelholm M, Hu G, Johnson WD, Kuriyan R, Kurpad A, Lambert EV, Maher C, Maia J, Matsudo V, Olds T, Onywera V, Sarmiento OL, Standage M, Tremblay MS, Tudor-Locke C, Zhao P, Church TS. The International Study of Childhood Obesity, Lifestyle and the Environment (ISCOLE): design and methods. BMC Public Health. 2013 Sep 30;13:900. doi: 10.1186/1471-2458-13-900. PMID 24079373
- [Result] Tudor-Locke C, Barreira TV, Schuna JM Jr, Mire EF, Katzmarzyk PT. Fully automated waist-worn accelerometer algorithm for detecting children's sleep-period time separate from 24-h physical activity or sedentary behaviors. Appl Physiol Nutr Metab. 2014 Jan;39(1):53-7. doi: 10.1139/apnm-2013-0173. Epub 2013 Jun 26. PMID 24383507
- [Result] Barreira TV, Schuna JM Jr, Mire EF, Katzmarzyk PT, Chaput JP, Leduc G, Tudor-Locke C. Identifying children's nocturnal sleep using 24-h waist accelerometry. Med Sci Sports Exerc. 2015 May;47(5):937-43. doi: 10.1249/MSS.0000000000000486. PMID 25202840
- [Result] Katzmarzyk PT, Barreira TV, Broyles ST, Champagne CM, Chaput JP, Fogelholm M, Hu G, Johnson WD, Kuriyan R, Kurpad A, Lambert EV, Maher C, Maia J, Matsudo V, Olds T, Onywera V, Sarmiento OL, Standage M, Tremblay MS, Tudor-Locke C, Zhao P, Church TS. Physical Activity, Sedentary Time, and Obesity in an International Sample of Children. Med Sci Sports Exerc. 2015 Oct;47(10):2062-9. doi: 10.1249/MSS.0000000000000649. PMID 25751770
- [Result] Tudor-Locke C, Barreira TV, Schuna JM Jr, Mire EF, Chaput JP, Fogelholm M, Hu G, Kuriyan R, Kurpad A, Lambert EV, Maher C, Maia J, Matsudo V, Olds T, Onywera V, Sarmiento OL, Standage M, Tremblay MS, Zhao P, Church TS, Katzmarzyk PT; ISCOLE Research Group. Improving wear time compliance with a 24-hour waist-worn accelerometer protocol in the International Study of Childhood Obesity, Lifestyle and the Environment (ISCOLE). Int J Behav Nutr Phys Act. 2015 Feb 11;12:11. doi: 10.1186/s12966-015-0172-x. PMID 25881074
- [Result] Pereira S, Gomes TN, Borges A, Santos D, Souza M, dos Santos FK, Chaves RN, Katzmarzyk PT, Maia JA. Variability and Stability in Daily Moderate-to-Vigorous Physical Activity among 10 Year Old Children. Int J Environ Res Public Health. 2015 Aug 7;12(8):9248-63. doi: 10.3390/ijerph120809248. PMID 26262632
- [Result] Gomes TN, Hedeker D, dos Santos FK, Pereira S, Katzmarzyk PT, Maia JA. Why Are Children Different in Their Daily Sedentariness? An Approach Based on the Mixed-Effects Location Scale Model. PLoS One. 2015 Jul 31;10(7):e0132192. doi: 10.1371/journal.pone.0132192. eCollection 2015. PMID 26230652
- [Result] Gomes TN, Katzmarzyk PT, dos Santos FK, de Chaves RN, Santos D, Pereira S, Champagne CM, Hedeker D, Maia J. Are BMI and Sedentariness Correlated? A Multilevel Study in Children. Nutrients. 2015 Jul 16;7(7):5889-904. doi: 10.3390/nu7075258. PMID 26193311
- [Result] Katzmarzyk PT, Barreira TV, Broyles ST, Champagne CM, Chaput JP, Fogelholm M, Hu G, Johnson WD, Kuriyan R, Kurpad A, Lambert EV, Maher C, Maia J, Matsudo V, Olds T, Onywera V, Sarmiento OL, Standage M, Tremblay MS, Tudor-Locke C, Zhao P, Church TS; ISCOLE Research Group. Relationship between lifestyle behaviors and obesity in children ages 9-11: Results from a 12-country study. Obesity (Silver Spring). 2015 Aug;23(8):1696-702. doi: 10.1002/oby.21152. Epub 2015 Jul 14. PMID 26173093
- [Result] LeBlanc AG, Katzmarzyk PT, Barreira TV, Broyles ST, Chaput JP, Church TS, Fogelholm M, Harrington DM, Hu G, Kuriyan R, Kurpad A, Lambert EV, Maher C, Maia J, Matsudo V, Olds T, Onywera V, Sarmiento OL, Standage M, Tudor-Locke C, Zhao P, Tremblay MS; ISCOLE Research Group. Correlates of Total Sedentary Time and Screen Time in 9-11 Year-Old Children around the World: The International Study of Childhood Obesity, Lifestyle and the Environment. PLoS One. 2015 Jun 11;10(6):e0129622. doi: 10.1371/journal.pone.0129622. eCollection 2015. PMID 26068231
- [Result] Pereira S, Katzmarzyk PT, Gomes TN, Borges A, Santos D, Souza M, dos Santos FK, Chaves RN, Champagne CM, Barreira TV, Maia JA. Profiling physical activity, diet, screen and sleep habits in Portuguese children. Nutrients. 2015 Jun 2;7(6):4345-62. doi: 10.3390/nu7064345. PMID 26043034
- [Result] Borghese MM, Tremblay MS, Katzmarzyk PT, Tudor-Locke C, Schuna JM Jr, Leduc G, Boyer C, LeBlanc AG, Chaput JP. Mediating role of television time, diet patterns, physical activity and sleep duration in the association between television in the bedroom and adiposity in 10 year-old children. Int J Behav Nutr Phys Act. 2015 May 13;12:60. doi: 10.1186/s12966-015-0221-5. PMID 25967920
- [Result] Tudor-Locke C, Mire EF, Dentro KN, Barreira TV, Schuna JM Jr, Zhao P, Tremblay MS, Standage M, Sarmiento OL, Onywera V, Olds T, Matsudo V, Maia J, Maher C, Lambert EV, Kurpad A, Kuriyan R, Hu G, Fogelholm M, Chaput JP, Church TS, Katzmarzyk PT; ISCOLE Research Group. A model for presenting accelerometer paradata in large studies: ISCOLE. Int J Behav Nutr Phys Act. 2015 Apr 20;12:52. doi: 10.1186/s12966-015-0213-5. PMID 25927615
- [Result] Ferrari GL, Oliveira LC, Araujo TL, Matsudo V, Barreira TV, Tudor-Locke C, Katzmarzyk P. Moderate-to-Vigorous Physical Activity and Sedentary Behavior: Independent Associations With Body Composition Variables in Brazilian Children. Pediatr Exerc Sci. 2015 Aug;27(3):380-9. doi: 10.1123/pes.2014-0150. Epub 2015 Apr 22. PMID 25902556
- [Result] Ferrari GL, Araujo TL, Oliveira L, Matsudo V, Mire E, Barreira TV, Tudor-Locke C, Katzmarzyk PT. Association Between Television Viewing and Physical Activity in 10-Year-Old Brazilian Children. J Phys Act Health. 2015 Oct;12(10):1401-8. doi: 10.1123/jpah.2014-0406. Epub 2015 Mar 31. PMID 25831554
- [Result] Borges A, Gomes TN, Santos D, Pereira S, dos Santos FK, Chaves R, Katzmarzyk PT, Maia J. A count model to study the correlates of 60 min of daily physical activity in Portuguese children. Int J Environ Res Public Health. 2015 Feb 26;12(3):2557-73. doi: 10.3390/ijerph120302557. PMID 25730296
- [Result] Gomes TN, Katzmarzyk PT, dos Santos FK, Souza M, Pereira S, Maia JA. Overweight and obesity in Portuguese children: prevalence and correlates. Int J Environ Res Public Health. 2014 Nov 3;11(11):11398-417. doi: 10.3390/ijerph111111398. PMID 25372884
- [Result] Gomes TN, dos Santos FK, Santos D, Pereira S, Chaves R, Katzmarzyk PT, Maia J. Correlates of sedentary time in children: a multilevel modelling approach. BMC Public Health. 2014 Aug 30;14:890. doi: 10.1186/1471-2458-14-890. PMID 25174736
- [Result] Muthuri SK, Wachira LJ, Onywera VO, Tremblay MS. Associations Between Parental Perceptions of the Neighborhood Environment and Childhood Physical Activity: Results from ISCOLE-Kenya. J Phys Act Health. 2016 Mar;13(3):333-43. doi: 10.1123/jpah.2014-0595. Epub 2015 Aug 13. PMID 26285040
- [Result] Borghese MM, Tremblay MS, Leduc G, Boyer C, Belanger P, LeBlanc AG, Francis C, Chaput JP. Television viewing and food intake during television viewing in normal-weight, overweight and obese 9- to 11-year-old Canadian children: a cross-sectional analysis. J Nutr Sci. 2015 Feb 27;4:e8. doi: 10.1017/jns.2014.72. eCollection 2015. PMID 26090104
- [Result] LeBlanc AG, Broyles ST, Chaput JP, Leduc G, Boyer C, Borghese MM, Tremblay MS. Correlates of objectively measured sedentary time and self-reported screen time in Canadian children. Int J Behav Nutr Phys Act. 2015 Mar 18;12:38. doi: 10.1186/s12966-015-0197-1. PMID 25889903
- [Result] Mcneil J, Tremblay MS, Leduc G, Boyer C, Belanger P, Leblanc AG, Borghese MM, Chaput JP. Objectively-measured sleep and its association with adiposity and physical activity in a sample of Canadian children. J Sleep Res. 2015 Apr;24(2):131-9. doi: 10.1111/jsr.12241. Epub 2014 Sep 30. PMID 25266575
- [Result] Chaput JP, Leduc G, Boyer C, Belanger P, LeBlanc AG, Borghese MM, Tremblay MS. Electronic screens in children's bedrooms and adiposity, physical activity and sleep: do the number and type of electronic devices matter? Can J Public Health. 2014 Jul 11;105(4):e273-9. doi: 10.17269/cjph.105.4511. PMID 25166130
- [Result] Muthuri SK, Wachira LJ, Onywera VO, Tremblay MS. Direct and self-reported measures of physical activity and sedentary behaviours by weight status in school-aged children: results from ISCOLE-Kenya. Ann Hum Biol. 2015;42(3):237-45. doi: 10.3109/03014460.2014.932847. Epub 2014 Jul 15. PMID 25026181
- [Result] Borghese MM, Tremblay MS, Leduc G, Boyer C, Belanger P, LeBlanc AG, Francis C, Chaput JP. Independent and combined associations of total sedentary time and television viewing time with food intake patterns of 9- to 11-year-old Canadian children. Appl Physiol Nutr Metab. 2014 Aug;39(8):937-43. doi: 10.1139/apnm-2013-0551. Epub 2014 Mar 14. PMID 24892903
- [Result] Larouche R, Chaput JP, Leduc G, Boyer C, Belanger P, LeBlanc AG, Borghese MM, Tremblay MS. A cross-sectional examination of socio-demographic and school-level correlates of children's school travel mode in Ottawa, Canada. BMC Public Health. 2014 May 23;14:497. doi: 10.1186/1471-2458-14-497. PMID 24886211
- [Result] Muthuri SK, Wachira LJ, Onywera VO, Tremblay MS. Correlates of objectively measured overweight/obesity and physical activity in Kenyan school children: results from ISCOLE-Kenya. BMC Public Health. 2014 May 9;14:436. doi: 10.1186/1471-2458-14-436. PMID 24885924
- [Derived] Santos MD, Ferrari G, Drenowatz C, Estivaleti JM, de Victo ER, de Oliveira LC, Matsudo V. Association between breastfeeding, parents' body mass index and birth weight with obesity indicators in children. BMC Pediatr. 2022 Oct 18;22(1):604. doi: 10.1186/s12887-022-03641-3. PMID 36258166
- [Derived] Barreira TV, Broyles ST, Tudor-Locke C, Chaput JP, Fogelholm M, Hu G, Kuriyan R, Lambert EV, Maher CA, Maia JA, Olds T, Onywera V, Sarmiento OL, Standage M, Tremblay MS, Katzmarzyk PT; ISCOLE Research Group. Epidemiological Transition in Physical Activity and Sedentary Time in Children. J Phys Act Health. 2019 Jun 27;16(7):518-524. doi: 10.1123/jpah.2018-0546. PMID 31104544
- [Derived] Zakrzewski-Fruer JK, Gillison FB, Katzmarzyk PT, Mire EF, Broyles ST, Champagne CM, Chaput JP, Denstel KD, Fogelholm M, Hu G, Lambert EV, Maher C, Maia J, Olds T, Onywera V, Sarmiento OL, Tremblay MS, Tudor-Locke C, Standage M; ISCOLE Research Group. Association between breakfast frequency and physical activity and sedentary time: a cross-sectional study in children from 12 countries. BMC Public Health. 2019 Feb 21;19(1):222. doi: 10.1186/s12889-019-6542-6. PMID 30791951
- [Derived] Wilkie HJ, Standage M, Gillison FB, Cumming SP, Katzmarzyk PT. Correlates of intensity-specific physical activity in children aged 9-11 years: a multilevel analysis of UK data from the International Study of Childhood Obesity, Lifestyle and the Environment. BMJ Open. 2018 Feb 3;8(2):e018373. doi: 10.1136/bmjopen-2017-018373. PMID 29431128
- [Derived] Sullivan SM, Broyles ST, Barreira TV, Chaput JP, Fogelholm M, Hu G, Kuriyan R, Kurpad A, Lambert EV, Maher C, Maia J, Matsudo V, Olds T, Onywera V, Sarmiento OL, Standage M, Tremblay MS, Tudor-Locke C, Zhao P, Katzmarzyk PT; ISCOLE Research Group. Associations of neighborhood social environment attributes and physical activity among 9-11 year old children from 12 countries. Health Place. 2017 Jul;46:183-191. doi: 10.1016/j.healthplace.2017.05.013. Epub 2017 May 22. PMID 28544991
- [Derived] Dumuid D, Olds T, Lewis LK, Martin-Fernandez JA, Katzmarzyk PT, Barreira T, Broyles ST, Chaput JP, Fogelholm M, Hu G, Kuriyan R, Kurpad A, Lambert EV, Maia J, Matsudo V, Onywera VO, Sarmiento OL, Standage M, Tremblay MS, Tudor-Locke C, Zhao P, Gillison F, Maher C; International Study of Childhood Obesity, Lifestyle and the Environment (ISCOLE) research group. Health-Related Quality of Life and Lifestyle Behavior Clusters in School-Aged Children from 12 Countries. J Pediatr. 2017 Apr;183:178-183.e2. doi: 10.1016/j.jpeds.2016.12.048. Epub 2017 Jan 10. PMID 28081885
- [Derived] Roman-Vinas B, Chaput JP, Katzmarzyk PT, Fogelholm M, Lambert EV, Maher C, Maia J, Olds T, Onywera V, Sarmiento OL, Standage M, Tudor-Locke C, Tremblay MS; ISCOLE Research Group. Proportion of children meeting recommendations for 24-hour movement guidelines and associations with adiposity in a 12-country study. Int J Behav Nutr Phys Act. 2016 Nov 25;13(1):123. doi: 10.1186/s12966-016-0449-8. PMID 27887654
- [Derived] Harrington DM, Gillison F, Broyles ST, Chaput JP, Fogelholm M, Hu G, Kuriyan R, Kurpad A, LeBlanc AG, Maher C, Maia J, Matsudo V, Olds T, Onywera V, Sarmiento OL, Standage M, Tremblay MS, Tudor-Locke C, Zhao P, Katzmarzyk PT; ISCOLE Research Group. Household-level correlates of children's physical activity levels in and across 12 countries. Obesity (Silver Spring). 2016 Oct;24(10):2150-7. doi: 10.1002/oby.21618. Epub 2016 Aug 25. PMID 27558527
- [Derived] Wilkie HJ, Standage M, Gillison FB, Cumming SP, Katzmarzyk PT. Multiple lifestyle behaviours and overweight and obesity among children aged 9-11 years: results from the UK site of the International Study of Childhood Obesity, Lifestyle and the Environment. BMJ Open. 2016 Feb 24;6(2):e010677. doi: 10.1136/bmjopen-2015-010677. PMID 26911589